CLINICAL TRIAL: NCT06141681
Title: Evaluation of Microcirculation With Photoplethysmography (Pulse Oximetry) in Healthy Volunteers and Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Principal Investigator, Nora Angélica Fuentes, Principal Investigator, Hospital Privado de Comunidad de Mar del Plata
Other Study IDs: UCI-000004
Record Dates: First submitted 2023-11-10; First posted 2023-11-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Microcirculation; Photoplethysmography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: >18 years old healthy
  Interventions: Other: photoplethysmography
- Patients in critical care unit: patient in ICU with requirement for hemodynamic monitoring
  Interventions: Other: photoplethysmography
- Patients with ventilatory support in the operating room or critical care unit: patient in the ICU or operating room with a requirement for hemodynamic monitoring and ventilatory support
  Interventions: Other: photoplethysmography

INTERVENTIONS:
Other: photoplethysmography — Photoplethysmography (BluePoint, Frankfurt, Germany) is the pulse wave measured by a pulse oximeter. It is obtained based on the absorbance of red/infrared light in a given tissue. The signal is made up of two components: 1) the alternating component (AC), which is the pulse wave itself, which is determined by the absorbance of pulsatile arterial blood. 2) The continuous component (DC), which represents the absorbance of venous blood and the rest of the tissues. Within these tests the investigators find vascular occlusion, elevation of the legs, raising or lowering the tested hand above/below the phlebostatic level, cold/heat test, etc. Each of them evaluates different aspects of circulation such as endothelial function, myogenic response to blood flow, perfusion pressure, autonomic reflexes, preload-dependence, or venous flow among other aspects of microcirculation.

SUMMARY:
The objective of this observational study is to explore microcirculation in healthy volunteers and in ventilated patients in the operating room and in critical care.

The general objective of this study is to evaluate microcirculation with photoplethysmography (PPG) in different pathophysiological situations and to compare PPG with available standard methods. Specifically, evaluate the correlation between the determinations of AC-DC waves obtained by Photoplethysmography (PPG) and those obtained in different dynamic tests in healthy volunteers.

To compare microcirculation assessments [capillary refill time (CRT), perfusion index (PI), perfusion index variability (PIV)] with measurements obtained by PPG in the context of critically ill patients.

To compare microcirculation assessments (CRT, PI PVI) with measurements obtained by PPG in the context of patients on invasive mechanical ventilation (IMV) in the operating room and in critical care.

DETAILED DESCRIPTION:
An attempt is made to explore different physiological aspects that affect microcirculation such as vascular tone and blood volume.

Photoplethysmography usually examines the AC wave equivalent to the pulsatile wave, however the DC component has been less explored and can account for the microcirculation and volemia status of the subjects.

Since there is no gold standard, it will be compared against different validated methods.

ELIGIBILITY:
Healthy Volunteers:

Inclusion Criteria:

* Written informed consent.
* Age > 18 years.

Exclusion Criteria:

* Pregnancy.
* Smokers.
* Respiratory and/or cardiovascular pathologies.
* Peripheral vascular disease.

Operation room or Critical care Unit patients

Inclusion criteria:

* Written informed consent.
* Age > 18 years.
* Critical patients ventilated in the ICU of any origin.

Exclusion criteria:

* Known peripheral vascular disease.
* Burns on both upper limbs.
* Trauma to both upper limbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers or operating room or intensive care patients- See inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
variations in AC signal of photoplethysmography | Through study completion, an average of 1 year
  Changes in the AC wave of photoplethysmography (it does not currently have standardized measurement units) will be evaluated in each functional test (CRT, LPR, venous occlusion test, progressive arterial occlusion test). It will be treated as a continuous numerical variable.
variations in DC signal of photoplethysmography | Through study completion, an average of 1 year
  Changes in the DC wave of photoplethysmography (it does not currently have standardized measurement units) will be evaluated in each functional test (CRT, LPR, venous occlusion test, progressive arterial occlusion test). It will be treated as a continuous numerical variable.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Fuentes, PhD, Principal Investigator — Hospital Privado de Comunidad
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina